CLINICAL TRIAL: NCT05852288
Title: Role of Inflammation in Carpal Tunnel Syndrome: A Prospective Cohort Study
Brief Title: Role of Inflammation in Carpal Tunnel Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/007075
Record Dates: First submitted 2023-04-19; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Carpal Tunnel Syndrome; Median Neuropathy, Carpal Tunnel
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with carpal tunnel syndrome: This study will follow a group of individuals with carpal tunnel syndrome (CTS) according to Bland's grading scale (grades 1-3) to assess the role of inflammation in CTS. Participants will undergo clinical and biochemical evaluations to assess inflammatory markers and CTS severity. The study will follow participants over time to determine the relationship between inflammation and CTS, which can inform the choice of transdermal drug administration.
  Interventions: Diagnostic Test: Inflammatory markers

INTERVENTIONS:
Diagnostic Test: Inflammatory markers — Participants in this cohort will undergo a comprehensive clinical and biochemical evaluation to assess the role of inflammation in CTS. The evaluation will include assessments of inflammatory markers, such as C-reactive protein (CRP), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α), as well as clinical measures of CTS severity.

SUMMARY:
This study aims to investigate the role of inflammation in carpal tunnel syndrome (CTS) using a prospective cohort study design. The study will involve a sample of at least 50 individuals with CTS who will undergo a comprehensive clinical and biochemical evaluation to assess the role of inflammation in CTS. The primary outcome measures include inflammatory markers, such as C-reactive protein (CRP), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α), as well as clinical measures of CTS severity. Data will be analyzed using regression analysis to determine the relationship between inflammation and CTS. The study is expected to provide information on the role of inflammation in CTS and inform the choice of drug and concentration for transdermal drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older
* Diagnosis of carpal tunnel syndrome based on clinical symptoms and nerve conduction studies
* Willingness and ability to provide informed consent to participate in the study
* Willingness and ability to comply with study procedures and follow-up visits

Exclusion Criteria:

* Presence of other neurological conditions that may affect nerve function in the upper extremities
* Use of medications that may affect inflammation or carpal tunnel syndrome severity
* History of previous carpal tunnel release surgery on the affected wrist
* Inability to comply with study procedures or follow-up visits
* Pregnancy or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will be recruited from a single center and will include at least 50 individuals with CTS. The population may include individuals of all ages, but the study will likely focus on middle-aged and older adults, as CTS is more common in this population.
  The study population will be diverse in terms of gender and race/ethnicity to ensure that the study findings are generalizable to a broader population.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
The relationship between inflammatory markers and symptom severity of carpal tunnel syndrome (CTS). | Changes of inflammatory markers and symptoms severity at baseline, 4 weeks, 8 weeks, and 12 weeks after baseline
  interleukin-6, tumor necrosis factor-alpha using blood tests. Symptom severity will be assessed with standardized questionnaire "the Boston Carpal Tunnel Questionnaire".
The relationship between inflammatory markers and grip strength of patients with CTS. | Changes of inflammatory markers and grip strength at baseline, 4 weeks, 8 weeks, and 12 weeks after baseline
  interleukin-6, tumor necrosis factor-alpha using blood tests. functional status by grip strength using a dynamometer.
The relationship between inflammatory markers and pinch strength of CTS patients. | Changes of inflammatory markers and pinch strength at baseline, 4 weeks, 8 weeks, and 12 weeks after baseline
  interleukin-6, tumor necrosis factor-alpha using blood tests. pinch strength will be measured using a dynamometer
The relationship between inflammatory markers and nerve conduction study of patients with CTS | Changes of inflammatory markers and nerve conduction study at baseline, 4 weeks, 8 weeks, and 12 weeks after baseline
  interleukin-6, tumor necrosis factor-alpha using blood tests. Nerve conduction study results (motor and sensory distal latency of median nerve and amplitude) will be used to determine CTS severity based on Bland's grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study will be available upon reasonable request. Requests for access to the data should be submitted via email to mohamed.elmeligie@acu.edu.eg. All requests will be reviewed by the study investigators to ensure that they are reasonable and consistent with the ethical principles of the study. Access to the data will be granted in compliance with applicable laws and regulations, and with appropriate safeguards to protect the privacy and confidentiality of study participants.
Supporting Information: SAP, ICF
Time Frame: After finishing the trial and up to 1 year.
Access Criteria: via email to mohamed.elmeligie@acu.edu.eg